CLINICAL TRIAL: NCT00220363
Title: A Phase 3, Parallel Group, Randomized, Double-Blind, Double-Dummy, Placebo and Active-Controlled Multicenter Trial to Investigate the Efficacy, Tolerability and Safety of Fesoterodine Sustained Release in Subjects With Overactive Bladder Syndrome
Brief Title: A Multicenter Trial to Investigate Fesoterodine Sustained Release in Overactive Bladder Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SP583
Record Dates: First submitted 2005-08-30; First posted 2005-09-22 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2008-04

CONDITIONS: Overactive Bladder Syndrome

INTERVENTIONS:
Drug: SPM 907

SUMMARY:
The trial consisted of a 2 week Run-In period, 12 week double-blind Treatment period and 2 week Safety Follow-Up period. Subjects were randomized to one of 4 treatment arms receiving either fesoterodine (SPM 907) 4mg, fesoterodine 8mg, active control (tolterodine SR 4mg) or placebo during the Double-Blind Treatment Period.

Two primary efficacy variables will be assessed for submission in the United States: change in the average number of micturitions (frequency) per 24 hours and the change in the average number of urge incontinence episodes per 24 hours. For the submissions in the European Union, the first primary variable will be the change in the average number of micturitions (frequency) per 24 hours and the co-primary variable is the treatment response, based on a treatment benefit scale. All continuous variables will be measured as changes from baseline to value after 12 weeks of treatment.

The most important safety variables included the assessment of adverse events, laboratory parameters, changes in ECG, physical exams and measurement of residual urine.

ELIGIBILITY:
Inclusion Criteria:

* Overactive Bladder Syndrome

Exclusion Criteria:

* less than 8 micturitions in 24 hours

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Axel Steinert, Study Director — UCB Pharma
Locations (1):
- Schwarz, Monheim, Germany

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Wagg AS, Herschorn S, Carlsson M, Fernet M, Oelke M. A plain language summary of the likelihood of symptom relief for patients taking fesoterodine for overactive bladder. J Comp Eff Res. 2022 Sep;11(13):919-925. doi: 10.2217/cer-2022-0041. Epub 2022 Jul 26. PMID 35881009
- [Derived] Cardozo L, Khullar V, El-Tahtawy A, Guan Z, Malhotra B, Staskin D. Modeling dose-response relationships of the effects of fesoterodine in patients with overactive bladder. BMC Urol. 2010 Aug 19;10:14. doi: 10.1186/1471-2490-10-14. PMID 20723260
- [Derived] Staskin D, Michel MC, Nitti V, Morrow JD, Wang J, Guan Z. Efficacy of fesoterodine over 24 hours in subjects with overactive bladder. Curr Med Res Opin. 2010 Apr;26(4):813-8. doi: 10.1185/03007990903585707. PMID 20121659